CLINICAL TRIAL: NCT00103337
Title: Phase II Evaluation of EMD121974 (NSC 707544, Cilengitide) in Asymptomatic Patients With Metastatic Androgen Independent Prostate Cancer
Brief Title: Cilengitide in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02904; UMCC 2004.030; N01CM62202 (NIH)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cilengitide

ARMS (2):
- Arm I (500 mg cilengitide) (Experimental): Patients receive lower dose cilengitide IV over 1 hour twice a week for 6 weeks.
  Interventions: Drug: cilengitide; Other: laboratory biomarker analysis
- Arm II (2000 mg cilengitide) (Experimental): Patients receive higher dose cilengitide IV over 1 hour twice a week for 6 weeks.
  Interventions: Drug: cilengitide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cilengitide — Given IV
  Other Names: EMD 121974
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well cilengitide works in treating patients with metastatic prostate cancer. Cilengitide may stop the growth of prostate cancer by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy, as measured by the rates of clinical progression at six-months, of two dose levels of EMD121974 in patients with asymptomatic metastatic androgen-independent prostate cancer.

SECONDARY OBJECTIVES:

I. To evaluate the safety of the two dose levels of EMD121974 in patients with metastatic androgen-independent prostate cancer.

II. To assess the objective response rate of two dose levels of EMD121974 in patients with metastatic androgen-independent prostate cancer and bidimensionally measurable disease.

III. To assess the rate of 50% or greater decline in the level of Prostate Specific Antigen.

TERTIARY OBJECTIVES:

I. To determine the effects of integrin αvβ3 and αvβ5 inhibition on total circulating tumor cells and endothelial cells isolated from peripheral blood and bone marrow aspirates from patients with metastatic androgen-independent prostate cancer.

II. To study the genotypic/phenotypic variances in circulating tumor cells in patients with metastatic androgen-independent prostate cancer before and after EMD121974 treatment.

III. To develop a genetic profile by cDNA microarray analysis of circulating tumor cells isolated from patients with metastatic androgen-independent prostate cancer before and after integrin αvβ3 and αvβ5 inhibition.

IV. Determine the effects of integrin αvβ3 and αvβ5 inhibition on systemic bone remodeling markers in patients with metastatic androgen-independent prostate cancer.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to prior bisphosphonate use (yes vs no). Patients are randomized to 1 of 2 doses of cilengitide.

ARM I: Patients receive lower dose cilengitide IV over 1 hour twice a week for 6 weeks.

AMR II: Patients receive higher dose cilengitide IV over 1 hour twice a week for 6 weeks.

In both arms, treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. After 2 courses, patients undergo response assessment. Patients achieving a complete response (CR) receive at least 3 additional courses beyond documentation of CR. Patients with partial response or stable disease continue treatment indefinitely in the absence of disease progression or unacceptable toxicity. Patients with a mixed response may continue treatment at the discretion of the investigator.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* A histologic or cytologic diagnosis of prostate cancer
* Metastatic disease that has progressed despite androgen deprivation therapy and antiandrogen withdrawal (28 days for flutamide and 42 days for bicalutamide or nilutamide); patients must demonstrate progression based on at least one of the following criteria:

  * Rising PSA - Defined as by one of the following criteria:

    * Three consecutive rising levels, with an interval of at least 2 weeks between each determination; the last determination must have a minimum value of >= 5 ng/ml and be determined within two weeks prior to registration
    * A PSA value of >= 20 ng/ml obtained within the 12 months prior to randomization and confirmed within 2 weeks prior to registration
    * A 50% rise in PSA values within 6 months prior to registration and confirmed within 2 weeks prior to registration; the last determination must have a minimum value of >= 5 ng/ml
  * Progression of bidimensionally measurable soft tissue (nodal metastasis) assessed within 28 days prior to registration by a CT scan or MRI of the abdomen and pelvis
  * Progression of bone disease (evaluable disease) (new bone lesion(s)) by bone scan within 42 days prior to registration
* ECOG performance status of 0-2
* Minimum PSA >= 5 ng/mL determined within 14 days of registration
* Testosterone < 50 ng/dL; patients must continue primary androgen deprivation with an LHRH analogue if they have not undergone orchiectomy
* Patients must have no prostate cancer-related pain, and no visceral metastasis (lung and/or liver)
* No prior chemotherapy for metastatic disease; no more than one prior non-cytotoxic therapy for metastatic disease
* No investigational or commercial agents or therapies may be administered with the intent to treat the patient's malignancy; four weeks must have elapsed since major surgery
* Prior radiotherapy is allowed as long as the bone marrow function is adequate
* Life expectancy of greater than 6 months
* WBC >= 3,000/µl
* ANC >= 1,500/µl
* Platelet count >= 100,000/µl
* Creatinine =< 1.5 x upper limits of normal
* Bilirubin within normal limits
* SGOT (AST) =< 2.5 x upper limits of normal
* SGPT (ALT) =< 2.5 x upper limits of normal
* The effects of EMD 121974 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because antiangiogenic agents are known to be teratogenic, men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document that is approved by the Institutional Human Investigation Committee (HIC)

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients may continue on a daily Multi-Vitamin, but all other herbal, alternative and food supplements (i.e. PC-Spes, Saw Palmetto, St John Wort, etc.) must be discontinued before registration
* Patients on stable doses of bisphosphonates which have been started no less than 6 weeks prior to protocol therapy, that show subsequent tumor progression, may continue on this medication, however patients are not allowed to initiate bisphosphonate therapy immediately prior or during the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not eligible; patients are not considered to have a "currently active" malignancy if they have completed therapy and are now considered without evidence of disease for 2 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical progression by bone scan or CT scan | 6 months

SECONDARY OUTCOMES:
Objective response using RECIST | Up to 30 days post-treatment
PSA response based on recommendations from the PSA Working Group | Up to 30 days post-treatment
Time to clinical response | Up to 30 days post-treatment
Time to PSA response | Up to 30 days post-treatment
Incidence of toxicity as assessed by CTCAE v3.0 | Up to 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, Principal Investigator — University of Michigan University Hospital
Locations (1):
- University of Michigan University Hospital, Ann Arbor, Michigan, United States